CLINICAL TRIAL: NCT04255407
Title: Evaluation of the Effect of Biophysical Stimulation With Pulsed Electromagnetic Fields on Intraspongious Bone Edema in Anterior Cruciate Ligament Reconstruction
Brief Title: Effect of Biophysical Stimulation on Intraspongious Bone Edema in Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEMF-LCA
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: ACL Injury; Pain; Magnetic Field Exposure
Keywords: bone bruise; pain; ACL reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Pain | interventions — Anti-Inflammatory Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-ONE® group (Experimental): I-ONE® therapy will be initiated in the 15 days preceding the ACL reconstruction surgery and in the first 60 days following the surgery.
  Paracetamol 1000 mg will be supplied to both groups, to be taken for pain control as per normal clinical practice.
  Interventions: Device: I-ONE® therapy
- Control group (Placebo Comparator): Patients will not be treated with I-ONE®. Pain will be treated with common NSAID and Paracetamol.
  Interventions: Drug: Anti-inflammatory drug

INTERVENTIONS:
Device: I-ONE® therapy — I-ONE® therapy will be used in patients with bone bruise on the knee after anterior cruciate ligament (ACL) injury 15 days before and 60 days after ACL reconstruction surgery for 4 hours a day compared to a control group (no-treatment).
  Other Names: I-ONE® IGEA
  Arms: I-ONE® group
Drug: Anti-inflammatory drug — Pain before and after ACL reconstruction will be managed with common anti-inflammatory drugs (Paracetamol)
  Arms: Control group

SUMMARY:
The following study has as main objective to evaluate whether the use of I-ONE® therapy can reduce post-operative pain thanks to the modulation of inflammation in patients with bone bruise on the knee after anterior cruciate ligament (ACL) injury if applied 15 days before and 60 days after ACL reconstruction surgery for 4 hours a day compared to a control group (no-treatment). Both groups will be able to take anti-inflammatory drugs for pain control as per normal clinical practice.

The secondary objective of the study are: quantify the reduction in the size of the bone bruise area, improving the level of knee function and the amount of anti-inflammatory drugs used in the aforementioned patients in the postoperative period compared to a control group.

DETAILED DESCRIPTION:
Articular cartilage, similarly to bone tissue, has a high sensitivity to physical stimuli and it has been shown that these are able to significantly modify the cartilage metabolism. There are several methods for applying a physical stimulus to articular cartilage: direct current, pulsed electromagnetic fields, electric fields and ultrasound. In vitro, all techniques have been shown to influence the metabolism of isolated chondrocytes. In vivo and in the clinic, the use of the biophysical stimulus for the treatment of the joint must respond to the need to treat the articular cartilage in its total extension and thickness, in addition to involving the joint structures, for example meniscus, ligaments, synovial membrane up to to the subchondral bone.

To date, these problems have been solved exclusively with the use of specific pulsed electromagnetic fields I-ONE®, as well demonstrated in the CRES study (Cartilage Repair and Electromagnetic Stimulation). In vitro, I-ONE® therapy produces a significant increase both in the proliferation of chondrocytes in the presence of Insulin growth factors- 1 (IGF-1), and in the synthesis of proteoglycans, also in the presence of inflammatory phenomena in the breeding ground, such as Interleukin 1B (IL-1B).

In vitro studies on neutrophils, synoviocytes and chondrocytes have shown that I-ONE® therapy increases the availability of adenosine A2A receptors and, acting as chondroprotective drugs, reduces tissue damage due to the inflammatory response. These results have been demonstrated in animal models of osteoarthritis where, stimulation with I-ONE® therapy led to a reduction in the progression of osteoarthritic knee injuries. In sheep undergoing osteochondral transplantation, I-ONE® therapy has been able to favor the formation of new subchondral tissue, decreasing the areas of resorption and avoiding its complete resorption. A high synthesis of anabolic factors, such as Transforming growth factor beta (TGF-β), and an inhibition of the synthesis of pro-inflammatory cytokines such as the Tumor necrosis factor alfa (TNF-α) and Interleukin 1 beta (IL-1β) have been observed as evidence of an anabolic and trophic effect. In rabbits subjected to osteochondral lesions, I-ONE® therapy has proven effective in significantly improving the quality of both bone and cartilage regenerated tissue in osteochondral defects in the presence of collagen scaffolds and Mesenchymal Stem Cells (MSCs). MSCs have the potential to differentiate into a chondrocyte phenotype however the presence of pro-inflammatory cytokines in particular IL-1β is able to inhibit chondrogenesis.

The anti-inflammatory activity of I-ONE® therapy effectively counteracted the degenerative effect of IL-1β by significantly improving cartilage regeneration compared to unstimulated lesions. This explains, even in vivo, the anti-degenerative, reparative and anti-inflammatory effect of treatment with I-ONE® therapy. In the clinical practice, I-ONE® therapy is able to prevent and/or slow down the degenerative phenomena that follow surgical operations. The latter result has been demonstrated both in patients undergoing anterior cruciate ligament reconstruction, and in patients with cartilage lesions treated with arthroscopic microfractures, in patients undergoing ONE STEP method with bone marrow concentrate and scaffold, and in patients undergoing total knee prosthesis with or without patellar resurfacing. All clinical studies have shown a reduction in NSAID intake and an anticipated functional recovery time in patients treated with I-ONE® therapy compared to those belonging to the non-treatment group. Also in the conservative treatment of joint pathologies, such as spontaneous osteonecrosis and knee osteoarthritis in the initial stagE I-ONE® therapy has proven effective in reducing the bone area marrow edema and in improving the functional recovery of the joint. Both in conservative and post-surgical treatment, the results were maintained even in the long term (follow-up 2 and 3 years after the treatment).

Similar results have been found after treatment with I-ONE® therapy in patients with patello-femoral pain, a frequent pathology in sports, especially in women, whose etiopathogenesis is controversial and attributable to several factors, including a malalignment of the joint, a dysplasia of the patella or of the femoral trochlea. The anterior knee pain, which accompanies this pathology, can become chronic over time and become highly limiting for sports. I-ONE® therapy has proven effective in promoting joint function, resolving painful symptoms and promoting a rapid return to sports, maintaining the result over a year. I-ONE® is an easy-to-use therapy that eliminates the possible side effects that characterize drug therapy and its use is well accepted by patients. Since cartilage degeneration is an irreversible process, it is essential to intervene early with an effective chondroprotective treatment, which is able to maintain an intact cartilage in the long run while also preserving the quality of the subchondral bone tissue (of fundamental importance for the survival of the articular cartilage).

In conclusion, the control of the joint microenvironment, by means of a non-invasive method, such as the biophysical stimulus, constitutes an important therapeutic possibility, which assumes a great importance in the presence of osteo-cartilaginous pain in the knee. In about 70% of the lesions of the anterior cruciate ligament (ACL), the presence of trabecular microfractures due to the impact of the subchondral bone, called bone bruises, is associated. These are characterized by the presence of hemorrhage, edema, necrosis and fibrosis: they are most frequently located in the external compartment of the knee (most often in the lateral femoral condyle) and associated with intense pain (accentuated by the weight-bearing). These lesions tend to reabsorb very slowly and cause intense pain especially during the post-operative period in ACL reconstruction, with limitation and lengthening of recovery times. This is mainly due to the difficulty of weight-bearing during the first post-operative month.

The following study has as main objective to evaluate whether the use of I-ONE® therapy can reduce post-operative pain thanks to the modulation of inflammation in patients with bone bruise on the knee after anterior cruciate ligament (ACL) injury if applied 15 days before and 60 days after ACL reconstruction surgery for 4 hours a day compared to a control group (no-treatment). Both groups will be able to take anti-inflammatory drugs for pain control as per normal clinical practice.

The secondary objective of the study are: quantify the reduction in the size of the bone bruise area, improving the level of knee function and the amount of anti-inflammatory drugs used in the aforementioned patients in the postoperative period compared to a control group.

I-ONE® therapy will be initiated in the 15 days preceding the ACL reconstruction surgery and in the first 60 days following the surgery, only in the treatment group. The control group will not be treated with I-ONE® devices (no-treatment). Paracetamol 1000 mg will be supplied to both groups, to be taken for pain control as per normal clinical practice.Drugs and I-ONE® devices will be delivered to the patient on the day of the pre-hospitalization visit which takes place routinely 15 days before the surgery. Clinical assessments using rating scales will be performed in both groups on the day of the pre-hospitalization visit, immediately before ACL reconstruction and during outpatient visit at 1, 2, 4, 12 and 24 months after ACL reconstruction. Magnetic resonance imaging will be performed 2, 4 and 12 months after surgery to highlight both the integration of the pro-ACL graft and the reduction of the bone bruise area. In particular, to quantify the resolution of the bone bruise area expected in the treatment group, the magnetic resonance performed 2 months after surgery will be used.

ELIGIBILITY:
Inclusion Criteria:

* patients completely sane and lucid
* acute lesion of the acl (date of trauma not exceeding 21 days)
* presence of bone bruise diagnosed by magnetic resonance imagine (diagnosed as presence of a hyperintense signal area at the subchondral bone level in the fast spin echo T2 scans with fat saturation or STIR (short tau inversion recovery)

Exclusion Criteria:

* patients who have undergone previous surgery on the same knee or lower limb
* patients with previous cartilage lesions of the affected knee
* patients with major axial deviations of the knee (varus or valgus alignment > 10°)
* patients who are taking cortisone therapies, use steroids, abuse alcohol
* menopausal women
* obesity (BMI> 30 Kg / m²)
* ongoing infections
* patients with rheumatoid arthritis, autoimmune diseases, systemic diseases, neoplasms
* reduced motility of the knee (active flexion equal or less than 90 ° before surgery)
* chronic rupture of the ACL (due to an injury of more than 21 days)
* 3rd grade medial collateral ligament rupture
* Grade 3 or 4 osteonecrosis according to the International Cartilage Repair Society (ICRS) classification criteria
* previous total meniscectomy

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 24 months
  It is a straight line with one end (scorse 0) meaning no pain and the other end (score 10) meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels.
Objective evaluation of the International Knee Documentation Committee | 24 months
  The International Knee Documentation Committee (IKDC Questionnaire) is a knee-specific patient-reported outcome which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). It's considered to be one of the most reliable outcome reporting tools in its category and was one of the instruments used in the popular MOON study. IKDC has been subjected to rigorous statistical evaluation and has proven to be a valid and responsive patient-reported outcome measure (PROM).
  Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Level of Tegner activity | 24 months
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer
Whole-Organ Magnetic Resonance Imaging Score (WORMS) of the knee in osteoarthritis. | 24 months
  To quantify the reduction of the area affected by bone edema, a semi-quantitative scoring method for multi-feature, whole-organ evaluation of the knee in osteoarthritis (OA) based on magnetic resonance imaging (MRI) findings will be used. Subarticular bone marrow abnormality was defined as poorly marginated areas of increased signal intensity in the normally fatty epiphyseal marrow on fat-suppressed T2-weighted FSE images. It will be evaluated in 15 different regions subdivided by anatomical landmarks in the fully extended knee and was graded from 0 to 3 based on the extent of regional involvement: 0=none; 1=<25% of the region; 2=25% to 50% of the region; 3=>50% of the region.
Monitoring of the intake of anti-inflammatory drugs | 24 months
  Patients will record in a diary all daily anti-inflammatory drug intake

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Zaffagnini, MD, PhD, Principal Investigator — IRCCS Istituto Ortopedico Rizzoli
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Papalia R, Torre G, Vasta S, Zampogna B, Pedersen DR, Denaro V, Amendola A. Bone bruises in anterior cruciate ligament injured knee and long-term outcomes. A review of the evidence. Open Access J Sports Med. 2015 Feb 18;6:37-48. doi: 10.2147/OAJSM.S75345. eCollection 2015. PMID 25733936
- [Result] Massari L, Benazzo F, De Mattei M, Setti S, Fini M; CRES Study Group. Effects of electrical physical stimuli on articular cartilage. J Bone Joint Surg Am. 2007 Oct;89 Suppl 3:152-61. doi: 10.2106/JBJS.G.00581. No abstract available. PMID 17908881
- [Result] Zorzi C, Dall'Oca C, Cadossi R, Setti S. Effects of pulsed electromagnetic fields on patients' recovery after arthroscopic surgery: prospective, randomized and double-blind study. Knee Surg Sports Traumatol Arthrosc. 2007 Jul;15(7):830-4. doi: 10.1007/s00167-007-0298-8. Epub 2007 Feb 28. PMID 17333120
- [Result] Moretti B, Notarnicola A, Moretti L, Setti S, De Terlizzi F, Pesce V, Patella V. I-ONE therapy in patients undergoing total knee arthroplasty: a prospective, randomized and controlled study. BMC Musculoskelet Disord. 2012 Jun 6;13:88. doi: 10.1186/1471-2474-13-88. PMID 22672794
- [Result] Adravanti P, Nicoletti S, Setti S, Ampollini A, de Girolamo L. Effect of pulsed electromagnetic field therapy in patients undergoing total knee arthroplasty: a randomised controlled trial. Int Orthop. 2014 Feb;38(2):397-403. doi: 10.1007/s00264-013-2216-7. Epub 2013 Dec 20. PMID 24352823